CLINICAL TRIAL: NCT03916068
Title: A Pilot Study Comparing Acute Post-Radiation Hyperbaric Oxygen (HBO2) Versus Trental and Vitamin E for Breast Cancer Patients Who Have Recently Completed Radiation Therapy as Part of Their Treatment Course
Brief Title: Acute Post-Radiation Hyperbaric Oxygen (HBO2) for Breast Cancer Patients Who Have Recently Completed Radiation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Legacy Health System (Other)
Responsible Party: Principal Investigator, Enoch Huang, Principal Investigator, Legacy Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HBO001
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Hyperbaric Oxygenation; Pentoxifylline; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyperbaric Oxygen Therapy (Experimental): Hyperbaric oxygen (HBO2) - 100% oxygen at 2.4 atmospheres ATA for 90 minutes, Monday-Friday for 30 sessions (six weeks)
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- Trental and Vitamin E (Active Comparator): Trental (pentoxifylline), 400 milligrams three times a day in combination with Vitamin E, 400 international units orally twice daily for six months
  Interventions: Drug: Trental Pill; Dietary Supplement: Vitamin E

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — Hyperbaric oxygen therapy at 2.4 atmospheres for 90 minutes for 30 sessions.
  Arms: Hyperbaric Oxygen Therapy
Drug: Trental Pill — Trental 400 mg three times daily, in combination with Vitamin E 400 IU twice daily
  Other Names: pentoxifylline
  Arms: Trental and Vitamin E
Dietary Supplement: Vitamin E — Vitamin E 400 IU twice daily, in combination with Trental 400 mg three times daily
  Arms: Trental and Vitamin E

SUMMARY:
This study aims to compare patients that receive hyperbaric oxygen or Trental and Vitamin E immediately after completion of radiation therapy to evaluate which treatment best reduces radiation fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Patient is currently undergoing treatment for breast cancer and is on one of two pathways:

  * Pathway 1 involves lumpectomy with radiation therapy, recurrence years later, mastectomy and tissue expander with further radiation therapy
  * Pathway 2 involves mastectomy and tissue expander, 6 weeks of radiation therapy, and an implant in 6 months
* Undergone mastectomy with expander or implant reconstruction > 2 weeks before starting radiation therapy
* Completed chest wall irradiation in the past 3 days
* Willing to stop herbal medications as directed by provider
* Willing to stop daily use of supplemental vitamin E (Multivitamin with vitamin E component is acceptable, vitamin E cream is also acceptable)
* Willing to have photographs of chest area taken for research purposes only
* Therapeutic PT-INR for participants taking Coumadin
* If tissue expanders remain intact during radiation, plan for conversion to the final implants must occur > 4 months after completing radiation
* Willing to travel to a Legacy Health facility for study related visits
* Agree to attend study visits outside of standard of care visits, if needed
* Willing to engage in pre/post testing and survey/phone calls
* Willing to attend all 6 weeks of HBOT if randomized to that group

Exclusion Criteria:

* < 18 years of age
* Pregnant or lactating
* Have final implant placed < 2 weeks before start of radiation therapy
* Plan to place final impacts < 4 months from the completion of radiation therapy, if tissue expanders are intact during radiation therapy
* Have evidence of ongoing infection or implant exposure before start of radiation therapy
* Radiation completed more than 3 days prior to study start
* Unable to comply with protocol
* Unable to provide written informed consent
* Unwilling or unable to stop oral supplemental Vitamin E
* PT-INR outside of acceptable range for participants taking Coumadin
* Any delay in radiation treatment greater than 14 days
* Investigator does not believe study participation is in the best interest of the patient
* History of a seizure within the last 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Change in breast fibrosis using Bakers Grade Assessment | Administered at week 1, week 7, week 13, week 25, week 53, and week 157.
  The Bakers Grade Assessment will be used to evaluate if lower incidence and severity of radiation fibrosis is observed in patients receiving post-operative hyperbaric oxygen treatment as compared to Trental and Vitamin E. The difference-from-baseline (DFB) score will be calculated to determine the incidence and severity of radiation fibrosis. Some patients may develop radiation fibrosis at a later time so the assessment will be done multiple throughout the three years to capture timing of fibrosis onset.

SECONDARY OUTCOMES:
Objective measurements of tissue pliability using a Tissue Compliance Meter | Obtained at week 1, week 7, week 13, week 25, week 53, and week 157.
Patients' sense of well-being using SF-20 Quality of life survey. | Administered at week 1, week 7, week 13, week 25, week 53, and week 157.
  Short Form 20 is a survey that patients complete to indicate their overall quality of life. The SF-20 is weighted and summed to provide easily interpretable scales for physical and mental health.
Pain in radiated breasts using a Visual Analog Scale | Administered at week 1, week 7, week 13, week 25, week 53, and week 157.
  Visual Analog Scale is a way for patients to assess their pain, on a scale of one to ten with ten being worst pain imaginable.
Presence of delayed wound healing, surgical complications, implant revision or loss | Evaluated at week 1, week 7, week 13, week 25, week 53, and week 157.

CONTACTS AND LOCATIONS:
Overall Officials: Enoch Huang, MD, Principal Investigator — Legacy Health System
Locations (1):
- Legacy Emanuel Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No